CLINICAL TRIAL: NCT03783468
Title: Early LIght Sedation Pressure Support in ARDS Patients
Brief Title: LIght Sedation Pressure Support
Acronym: LIPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decision
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_18; 2018-A01036-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-11; First posted 2018-12-21 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- light sedation pressure support ventilation (Experimental)
  Interventions: Other: decrease of sedation doses and switch of ventilator settings

INTERVENTIONS:
Other: decrease of sedation doses and switch of ventilator settings — tapering sedation doses (propofol) switch from assisted ventilation to pressure support ventilation

SUMMARY:
Sedation may have many drawbacks in ICU patients: cardiovascular, neurologic, muscular.

Light sedation and Pressure Support ventilation is feasible in ARDS patients. However spontaneous breathing can lead to high transpulmonary pressure.

The goal of the study is to measure transpulmonary pressure before sedation decrease and after stabilization. The main endpoint is transpulmonary pressure less than 24 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* ARDS (Berlin definition)
* social insurance

Exclusion Criteria:

* neuromuscular disorders
* pregnancy
* need for muscular paralysis
* need for deep neurosedation
* more than 24hrs of artificial ventilation
* cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
transpulmonary pressure at early stabilization of patient | when patient is conscious and stable (no modification of ventilator settings) generally within 2 hours
  transpulmonary pressure (Paw - Peso < 24 cmH2O)

SECONDARY OUTCOMES:
oxygenation modification | stabilization of ventilator settings; 1hour after stabilization of ventilator settings
  PaO2/FiO2
arterial pressure modification | stabilization of ventilator settings; 1hour after stabilization of ventilator settings
  Mean arterial pressure
Heart rate modification | stabilization of ventilator settings;1hour after stabilization of ventilator settings
  heart rate
vasopressor dose modification | stabilization of ventilator settings ; 1hour after stabilization of ventilator settings
  vasopressor dose in norepinephrine equivalent
acquired neuromyopathy | ICU discharge, an average 16 days
  MRC <48/60
muscular volume decrease | at 24 hours; at day of extubation; ICU discharge, an average 16 days
  quadriceps volume assessed by echography
ventilator free days | during the first 28 days
  ventilator free days until day 28
delirium in ICU | ICU discharge, an average 16 days
  CAM-ICU is a valid and reliable delirium assessment tool recommended by the Society of Critical Care Medicine (SCCM) in its 2013 Pain, Agitation and Delirium (PAD) guidelines. the presence of delirium is confirmed in the presence of criteria 1, 2 and 3 or 4.
change of the functional respiratory parameters from baseline at 6 months | at 6 months
  vital capacity, total pulmonary capacity,
PTSD | at 6 months
  post traumatic stress disorder impact of event scale > 33 tems are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely") and the total score (ranging from 0 to 88)
number of auto extubation | whatever until ICU discharge, an average 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Ledoux, MD, Principal Investigator — University Hospital, Lille